CLINICAL TRIAL: NCT03346161
Title: Optimizing Decision Making About Breast Reconstruction After Mastectomy: A Patient-Centered Approach
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201701045
Record Dates: First submitted 2017-11-01; First posted 2017-11-17 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Demography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: BREASTChoice (Decision Tool) (Experimental): Investigators recruited patients scheduled for a plastic/reconstruction consult. Investigators identified patients who completed a mastectomy, or were scheduled for one, and considering reconstruction, but didn't have an appointment with a plastic/reconstructive surgeon. A study team member called the patient to determine their interest and offered for them to come to their scheduled appointment 30 minutes early to meet a coordinator or offered them the option to complete pre-appointment procedures at home. Patients randomized using computer random assignment. If the patient didn't have an appointment, she scheduled a convenient time to complete study procedures with research staff. Patients interacted with the decision tool. They were asked to answer a survey. After the appointment, the team collected information consult duration, decision process quality, and measures of shared decision making. Patient participation was approximately 30 minutes.
  Interventions: Other: Decision tool; Other: Decision Group - Outcome Measures; Other: Demographic and Background Questions
- Arm 2: Enhanced Usual Care (Surgical Care Booklet) (Active Comparator): Investigators recruited patients scheduled for plastic/reconstruction consultation. Investigators identified patients who completed or scheduled a mastectomy, and considering reconstruction, but didn't have an appointment with a plastic/reconstructive surgeon. A study team member called the patient to determine their interest and offered for them to come to their scheduled appointment 30 minutes early to meet a coordinator or to complete the pre-appointment procedures at home. Patients were randomized using computer random assignment. If the patient didn't have an appointment, she scheduled a convenient time to complete study procedures with research staff. Patients interacted with American Society of Plastic Surgeons booklet "Breast Reconstruction." They were asked to answer a survey. After the appointment, the team collected information about consult duration, decision process quality, and measures of shared decision making. Patient participation was approximately 30 minutes.
  Interventions: Other: Usual care American Society of Plastic Surgeons booklet "Breast Reconstruction"; Other: Usual Care Group - Outcome Measures; Other: Demographic and Background Questions

INTERVENTIONS:
Other: Usual care American Society of Plastic Surgeons booklet "Breast Reconstruction" — -Booklet from the American Society of Plastic Surgeons about how to choose a breast reconstruction surgeon, what to expect during surgery, what is breast reconstruction, risks of breast reconstruction, recovery, costs, and questions to ask surgeon about breast reconstruction
  Arms: Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Other: Decision tool — -Interactive web based tool. Provides detail about breast reconstruction, asks participant questions about health and medications to personalize risks for breast reconstruction outcome. The tool also goes into pros/cons of breast reconstruction, talks about differences between types of reconstruction, helps people weigh when to have reconstruction (immediate vs. delayed), shows participants representative photos of breast reconstruction outcomes, and assesses patients' knowledge and preferences
  Arms: Arm 1: BREASTChoice (Decision Tool)
Other: Usual Care Group - Outcome Measures — * Section 1 Knowledge (primary outcome) - set of multiple choice questions about breast reconstruction, implants, flap surgeries, and side effects
  * Section 2 Decisional Conflict Scale - 4 questions with yes/no answers dealing with participant's certainty about surgery (it total score less than 4, indicates higher decisional conflict)
  * Section 3 Patient Activation Measures: 3 yes/no questions about participant's knowledge and trust of healthcare provider, sources of info about breast reconstruction, and different options available
  * Section 4 Breast Reconstruction Decision Quality Instrument: 18 multiple choice questions about thought and processes that went into deciding about breast reconstruction
  * Section 5 BREAST-Q: 3 questions about the breast reconstruction consultation appoint answers range from 0=no effort to 9=every effort.
  Arms: Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Other: Decision Group - Outcome Measures — * Section 1 Knowledge and Values Clarification Questions - set of multiple choice questions about the participants feelings on breast reconstruction, implants, flap surgeries, and side effects
  * Section 2 Decisional Conflict SURE measure - 4 questions with yes/no answers dealing with participant's conflicts on surgery (if total score less than 4, indicates higher clinical significant decisional conflict)
  * Section 3 Patient Activation Measures: 3 yes/no questions about participant's knowledge and trust of healthcare provider, sources of info about breast reconstruction, and different options available
  * Section 4 Breast Reconstruction Decision Quality Instrument: 18 multiple choice questions about thought and processes that went into deciding about breast reconstruction (for those who have a clinical visit)
  * Section 5 BREAST-Q: 3 questions about the breast reconstruction consultation appointment answers range from 0=no effort to 9=every effort (for those who have a clinical visit).
  Arms: Arm 1: BREASTChoice (Decision Tool)
Other: Demographic and Background Questions — * Asks 15 questions
  * Age, education, ethnicity, race, combined household income, zip code, disease stage, (3) questions about health insurance, (4) questions about participant's ability to work with numbers, heath literacy, health insurance status, and (1) question on if participant spoke to another provider about breast reconstruction decision

SUMMARY:
Although clinical decision tools (CDTs) exist for a variety of treatments, CDTs designed to support personalized breast reconstruction decisions, particularly about type and timing of reconstruction, are lacking. The objective of this proposal is to develop and pilot test a clinical decision tool that provides personalized risk information and reflects patients' preferences and clinical needs.

ELIGIBILITY:
* Newly diagnosed or recurrent breast cancer
* Considering a referral or already referred to a plastic surgeon by their surgical oncologist for possible reconstruction
* Considering or completing a mastectomy.
* Does not have known distant metastatic disease (stage IV disease) at the time of recruitment
* Female.
* English-speaking.
* At least 18 years of age.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Myckatyn, M.D., Principal Investigator — Washington University School of Medicine; Mary C Politi, Ph.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to participant enrollment on 01/12/2018 and closed to participant enrollment on 10/24/2018.
Period: Overall Study
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet) | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Full Range); unit: years] | 52.3 [31 to 77] | 49.1 [25 to 74] | 50.7 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 56 | 58 | 114
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 6 | 9
  White | 49 | 52 | 101
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percent Correct on the Knowledge Measure (Objective Knowledge Score)
Description: To determine whether the CDT increases knowledge about their choice, the investigators will compare objective knowledge scores between participants using the CDT and those who received usual care
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: percentage of answers correct
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 60
percentage of answers correct | 84.6 (14.2) | 59.7 (18.0)

2. Primary Outcome: Decisional Conflict (SURE Measure)
Description: * To determine whether the CDT reduces uncertainty about choice. Participants are asked to report how sure they feel about their choice, if they have enough information to understand the choice, if they are clear about the risks and benefits, and if they have enough support to make a choice. Results are compared between the BREASTChoice and Enhanced Usual Care groups.
  * Higher SURE values indicate certainty in choice
  * Scores range from 0-4
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 60
score on a scale | 2.9 (1.2) | 2.5 (1.4)

3. Primary Outcome: Decision Process (Decision Quality Index Subscale)
Description: * The total points are summed and then divided by the total number of items to result in scores from 0-100%, with higher scores indicating a more shared decision making process
  * Assess the extent to which patients were meaningfully involved in decision-making with their clinicians
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 60
score on a scale | 65.1 (21.5) | 58.2 (20.7)

4. Secondary Outcome: Quality of Life as Measured by the BREAST-Q Questionnaire
Description: * Assessed 4 subscales: satisfaction with breasts, psychosocial well-being, physical well-being, and sexual well-being
  * Score from 0 (worst) to 100 (best). Higher scores reflect a better outcome.
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 60
score on a scale
  Satisfaction with breasts | 58.5 (24.8) | 57.3 (23.7)
  Psychosocial well-being | 64.6 (19.9) | 71.2 (17.6)
  Physical well-being | 79.5 (18.1) | 82.7 (16.5)
  Sexual well-being | 56.3 (19.4) | 61.2 (19.2)

5. Secondary Outcome: Gold Standard Shared Decision Making as Measured by the Top collaboRATE Score
Description: * Top collaboRATE score = the percentage of patients from whom there was 'gold standard' shared decision making as assessed by the collaboRATE measure
  * The top score is coded as '1', if the response to all three collaboRATE items was less than 9. Then the investigators calculated the percentage of all encounters that were coded as '1' indicating gold standard shared decision making.
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Population: 3 participants from Arm 1 were excluded from the outcome measure as their data was missing. 1 participants from Arm 2 was excluded from the outcome measure as her data was missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 56 | 59
Participants | 33 | 37

6. Secondary Outcome: Patient Activation (PAM) as Measured by the Number of Participants Who Agreed With Each Statement
Description: -3 questions consisting of the following:
  * I am confident I can tell my healthcare provider concerns that I have about breast reconstruction even when he or she does not ask (confidence in healthcare provider)
  * I am confident I can find trustworthy sources of information about my breast reconstruction decision (confidence in trustworthy sources)
  * I know the different options available for breast reconstruction (knowledge on breast reconstruction options)
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Population: 3 participants in the BREASTChoice arm did not provide an answer to this question and are not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 57 | 60
Participants
  Confidence in healthcare provider | 55 | 59
  Confidence in trustworthy sources | 57 | 58
  Knowledge on breast reconstruction options | 56 | 50

7. Secondary Outcome: Receipt of Reconstruction
Description: Assessed if participants received reconstruction
Time Frame: Through follow-up (approximately 6 months)
Population: 2 participants in the Enhanced Usual Care arm have not had their reconstruction surgery but are planning to schedule it but it is outside the follow-up window.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 58
Participants
  Yes | 48 | 47
  No/Not yet started | 11 | 8
  Not applicable (breast-conserving surgery) | 1 | 3

8. Secondary Outcome: Type of Reconstruction
Description: Assessed what type of reconstruction participants received
Time Frame: Through completion of follow-up (approximately 6 months)
Population: Only patients who had reconstruction are applicable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 48 | 47
Participants
  Implant | 23 | 27
  Flap | 10 | 8
  Unknown | 15 | 12

9. Secondary Outcome: Timing of Reconstruction
Description: * Assessed timing of reconstruction
  * Immediate is defined as reconstruction at the time of mastectomy
  * Delayed is defined as reconstruction any time after the mastectomy and performed as a separate surgery
Time Frame: Through completion of follow-up (approximately 6 months)
Population: Only patients who had reconstruction are applicable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 48 | 47
Participants
  Immediate | 45 | 47
  Delayed | 3 | 0

10. Secondary Outcome: Time Spent on Tool
Description: How long participants spent on the BREASTChoice tool
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Population: -Only patients randomized to BREASTChoice (Decision Tool) are evaluable for this outcome measure
Measure: Median (Full Range); unit: minutes
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 0
minutes | 26.7 [9.9 to 130.2] |

11. Secondary Outcome: Consult Time
Description: Assessed the time between when the plastic/reconstructive surgeon entered and exited the consult room (not including time spent with a resident, nurse, or other clinical staff)
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Measure: Mean (Full Range); unit: minutes
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 60
minutes | 29.9 [10 to 58] | 30 [9 to 65]

12. Secondary Outcome: Usability as Measured by the Computer System Usability Questionnaire (CSUQ)
Description: * Assessed ease of usability of the BREASTChoice tool
  * Scale is from 1 (strongly disagree) to 7 (strongly agree)
Time Frame: Through completion of breast consultation appointment (total participant time approximately 30 minutes)
Population: -Only patients randomized to BREASTChoice (Decision Tool) are evaluable for this outcome measure
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
Number analyzed (Participants) | 60 | 0
score on a scale | 6.3 [4.8 to 7.0] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of study enrollment until completion of patient follow-up (approximately 15 months)
Arm/Group | Arm 1: BREASTChoice (Decision Tool) | Arm 2: Enhanced Usual Care (Surgical Care Booklet)
All-Cause Mortality (participants affected / at risk) | 1/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03346161/Prot_SAP_000.pdf